CLINICAL TRIAL: NCT05577026
Title: Safe and Appropriate Prescribing of Opioids in Primary Care: a Randomized Control Trial
Brief Title: Safe Prescription of Opioids in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Smartaval2022-01
Record Dates: First submitted 2022-10-04; First posted 2022-10-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Opioid-Related Disorders; Narcotic-Related Disorders; Addiction
Keywords: Early Intervention, Educational; Prescription Drugs; Opioids; Primary Health Care
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Educational intervention with prescription feedback (Experimental): Healthcare personnel will participate in a brief educational intervention with information regarding treatment guidelines, recommendations, and risks of prescribing opioids. The presentation will include benchmarking on clinic opioid prescription patterns compared to other primary health centers, followed by targeted feedback on prescription patterns over the subsequent 12 months. Standardized materials will be provided, including a patient-provider agreement, outline of a patient treatment plan, and recommendations of how shared routines at the center can be improved.
  Interventions: Behavioral: Educational intervention and prescription feedback
- Written information on guidelines (Active Comparator): The manager at each PHC center in the active control group will receive written information on treatment guidelines for pain management. These centers will not receive the intervention, consisting of the onsite educational visit and targeted prescription feedback.
  Interventions: Behavioral: General information on treatment guidelines
- Standard care (No Intervention): The passive control group will consist of PHC centers that met the eligibility criteria for the study but did not actively participate in the study. Care as usual will proceed at the centers. Prescription data will be gathered directly from regional registers and databases; thus there will be no need to communicate directly with the centers. This arm will be used only if the General Data Protection Regulation continues to allow access to regional registers and databases in primary health care.

INTERVENTIONS:
Behavioral: Educational intervention and prescription feedback — Brief educational intervention and patient and provider materials regarding prescription of opioids. Subsequent feedback on clinic prescription of opioids over 12 months.
  Arms: Educational intervention with prescription feedback
Behavioral: General information on treatment guidelines — Written information on guidelines and recommendations regarding prescription of opioids.
  Arms: Written information on guidelines

SUMMARY:
Opioid analgesics are commonly prescribed addictive narcotics intended for the treatment of pain. Inappropriate prescription of opioids in quantities and for conditions which lack clinical evidence contributes to the risk of misuse and addiction. The majority of opioid prescriptions are written by physicians (general practitioners) in primary health care (PHC). PHC is thus an important setting for efforts to encourage the safe and appropriate prescription of opioids. Increasing knowledge of pain treatment recommendations, risks of opioids, and guidelines for the prescription of opioids may decrease inappropriate prescription, and thereby risk of tolerance, dependence, and addiction.

DETAILED DESCRIPTION:
Opioids are a class of addictive narcotic drugs which can be obtained by prescription for the treatment of pain. There is clinical evidence for the use of opioids for acute, post-operative, and cancer related pain, although guidelines recommend the lowest effective dose and duration be prescribed. There is less evidence for the long-term benefits of opioid therapy for chronic non-cancer pain and the risk for harm and addiction is increased with prolonged use. Patients with long-term treatment may experience only marginal pain reduction and a risk of long-term consequences including tolerance, dependence, and adverse effects such as cognitive disturbance and decline, behavioral problems, emergency visits, accidents, suicide, and drug-related mortality. As the majority of opioids are prescribed by physicians in primary health care, this is an important setting for promoting the safe and appropriate use of prescription opioids.

This trial evaluates whether a brief educational intervention in primary health care (PHC) followed by 12 months of feedback on prescription data changes the prescription of opioids in primary care.

PHC centers in Stockholm County will be invited to participate in the study. Centers that express interest in participating, meet the inclusion criteria, and do not meet the exclusion criteria will be randomized to the intervention or control group. Personnel at the intervention centers will participate in a brief educational intervention followed by 12 months of regular feedback on opioid prescriptions, with benchmarking to other local PHC centers. Centers randomized to the active control group will receive written information on treatment guidelines but will not receive the onsite educational intervention or prescription feedback.

The primary outcome, change in opioid prescription, will be measured at 12 months after intervention start. Data on outcomes and characteristics of participating primary health care centers including prescription before, during and after the intervention will be extracted from regional health care registers and databases and analyzed statistically.

ELIGIBILITY:
Eligibility criteria apply to primary health care centers.

Inclusion Criteria:

* Employs at least two full-time physicians
* Has at least 3000 listed patients
* Has a regional care agreement (contract)
* Connected to the regional quality register (Stockholm County)

Exclusion Criteria:

* In operation for less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in opioid prescriptions | 12 months
  Change in prescription of opioids as measured by defined daily dose (DDD)

SECONDARY OUTCOMES:
Change in opioid types | 12 months
  Change in type of opioids prescribed by drug class (ATC code)
Change in opioid prescriptions | 24 months
  Change in prescriptions of opioids as measured by defined daily dose (DDD)

OTHER OUTCOMES:
Change in number of patients with opioid prescriptions | 12 months
  Change in number of patients prescribed opioids (new or continued prescription)
Change in initial opioid prescriptions | 12 months
  Change in number of patients with initial (new) opioid prescriptions among opioid-naïve patients

CONTACTS AND LOCATIONS:
Overall Officials: Johan Franck, MD, PhD, Principal Investigator — Region Stockholm / SLSO
Locations (1):
- Akademiskt Primärvårdscentrum, Solnavägen 1D, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data for this study will be gathered from regional registers and health care databases. For permission to access these data, interested parties should contact Region Stockholm.

REFERENCES:
- [Derived] Kruger C, Franck J, Hallgren J, Af Winklerfelt Hammarberg S, Norman C, Niper A, Westman J. Improved opioid prescribing in primary care: protocol for a cluster randomised pragmatic trial. BMJ Open. 2025 Dec 17;15(12):e110818. doi: 10.1136/bmjopen-2025-110818. PMID 41407431